CLINICAL TRIAL: NCT06911086
Title: SH-LPS System in Preoperative Planning for Liver Resection: a Randomized Controlled Trial
Brief Title: SH-LPS System in Preoperative Planning for Liver Resection
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yuhua Zhang, MD, Principal Investigator, Director of Hepatopancreatobiliary Surgery, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2025-27（IIT）
Record Dates: First submitted 2025-03-05; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Liver Tumor; Surgery; 3D Printing; Preoperative Planning
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D group (Experimental): A three-dimensional digital model is constructed based on the patient's CT/MRI data and a physical model is printed. Using the model's self-healing property after cutting, multiple simulated surgeries are performed to help plan the optimal surgical approach. The best surgical path derived from the model is combined with traditional CT/MRI data to determine the final surgical path, and the surgery is then performed according to this finalized path.
  Interventions: Device: 3D printed models
- CT/MRI group (Sham Comparator): The surgical approach is planned based on traditional two-dimensional CT/MRI images, and the surgery is performed according to this planned path.
  Interventions: Other: CT or MRI image

INTERVENTIONS:
Device: 3D printed models — A three-dimensional digital model is constructed based on the patient's preoperative CT/MRI images, and a personalized physical model is created using 3D printing. This model has the ability to self-heal after being cut. Surgeons can perform multiple simulated surgeries on the model to plan the optimal surgical path before the authetic surgery
  Arms: 3D group
Other: CT or MRI image — Obtain the patient's CT/MRI images and determine the definitive surgical path based on the two-dimensional images.
  Arms: CT/MRI group

SUMMARY:
Effective preoperative planning and real-time intraoperative guidance are crucial for performing accurate liver resections. To address this need, the researchers have designed advanced 3D-printed liver models using a self-healing elastomer, created through the copolymerization of 4-acryloylmorpholine (ACMO) and methoxy poly(ethylene glycol) acrylate (mPEGA). These models demonstrate outstanding healing properties, swiftly restoring their structure within minutes at room temperature, and quickly recovering after incisions.

In previous studies, Professor Yuhua Zhang, the project applicant, collaborated with a team from Zhejiang University to develop a 3D-printed liver model that is self-healing and reusable for repeated cutting. They preliminarily explored the feasibility of applying this model for preoperative planning and surgical training for liver surgeries. The results were published in Nature Communications (Lu et al., Nat Commun. Dec 19;14(1):8447). Building on this, the applicant intends to establish a personalized liver surgery planning system (Personalized Liver Surgery Planning System Based on High-Fidelity 3D Printed Self-Healing Liver Models, SH-LPS), which will assess, through a randomized controlled trial, the value of SH-LPS in improving liver surgery efficiency and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* Patients with a resectable tumor in the liver;
* Eastern Cooperative Oncology Group Performance status score: 0;
* Child-Pugh classification: A;
* The Laboratory test results meet the following criteria and patients can tolerate surgery: Haemoglobin≥90g/L, Neutrophil count≥1.5×10⁹/L, Platelet count≥100×10⁹/L, Aspartate or alanine aminotransferase≤5 upper limits of normal(ULN）, alkaline phosphatase≤2.5 ULN, Serum albumin≥30g/L, serum creatinine<1.5 ULN, International normalized ratios（INR）≤2 or rothrombin time（PT）exceed ULN≤6s, Creatinine clearance≥60 mL/min.

Exclusion Criteria:

* Patients with extra-hepatic metastasis;
* Anti-cancer therapy or surgery such as radiotherapy, radiofrequency ablation in 28 days prior to the surgery;
* Clinically significant bleeding or bleeding tendencies within 3 months prior to enrollment or on thrombolytic or anticoagulant therapy;
* Severe lung disease (eg, acute lung disease, pulmonary fibrosis that affects lung function, interstitial lung disease), uncontrolled diabetes mellitus (fasting blood glucose ≥10 mmol/L);
* There are other unsuitable candidates for clinical trials, such as mental illness or alcohol dependence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Opertation duration | Until the end of the surgey
  The duration from the start to the end of the surgery.
Blood loss | Until the end of the surgey
  Blood loss during the operation

SECONDARY OUTCOMES:
R0 resection rate | Until the day the official pathology report comes out, an average of two weeks
  The percentage of surgical cases in which the tumor is completely removed with no microscopic residual cancer cells left at the margins of the resected tissue
Surgical complications | Until three months after the surgery
  The incidence rate of surgical complications
Postoperative hospital stay. | Until the day the patient is discharged, an average of one week.
  Postoperative hospital stay refers to the period of time a patient remains in the hospital after undergoing surgery, until they are medically stable and deemed fit for discharge.

IPD SHARING:
Plan to Share IPD: No